CLINICAL TRIAL: NCT05036265
Title: Laparoscopic Liver Resection for Colorectal Liver Metastases: Retrospective Analysis of Prognostic Factors and Oncological Outcomes in a Single-center Cohort
Brief Title: Prognostic Factors and Oncological Outcomes in Laparoscopic Liver Resection for CRLM
Status: Completed | Type: Observational
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Dr. M. D'hondt, Dr Mathieu D'Hondt, Principal Investigator, General Hospital Groeninge
Other Study IDs: B396201939301
Record Dates: First submitted 2021-08-23; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer; Liver Metastases; Surgery
Keywords: hepatopancreatobiliary; laparoscopic liver resection; colorectal liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Laparoscopic liver resection (LLR) has gained acceptance as an effective treatment for colorectal liver metastases (CRLM) in selected patients, providing similar oncologic outcomes compared to open liver resection (OLR). A single-center retrospective analysis of a prospectively maintained database was performed. The primary aim of this study was to determine prognostic factors for the survival outcomes associated with LLR for CRLM.

DETAILED DESCRIPTION:
LLR was defined as pure LLR, including conversions to OLR. In case of missing data, additional details were retrieved from the individual patient file. Data on patient demographics, timing of diagnosis, neoadjuvant chemotherapy (NAC), tumor characteristics (both primary tumor and CRLM), histopathology, molecular characteristics, operative technique (including classification into anatomically major/technically major/minor LR), intra- and postoperative course, adjuvant chemotherapy (AC) as well as oncological outcomes (OS and DFS) were gathered and analyzed. Postoperative complications were graded according to the Clavien-Dindo classification. Complications were classified as major in case of Clavien-Dindo ≥ 3A.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colorectal liver metastases
* Patients who received laparoscopic liver resection for colorectal liver metastases
* Patients who received the laparoscopic liver resection between September 2011 and mid-March 2020

Exclusion Criteria:

* Patients with contraindication for laparoscopic liver resection
* Refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received laparoscopic liver resection for colorectal liver metastases at General Hospital Groeninge between September 2011 and mid-March 2020
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Survival outcomes | 9 years
  Overall and disease-free survival (Kaplan-Meier method)
Prognostic factors | 9 years
  Univariate Cox proportional-hazards regression analysis